CLINICAL TRIAL: NCT07388979
Title: MAGIa In-vitro- Diagnostics Medical Device Dedicated to Combined Screening of HIV, HBV, HCV and Syphilis and HBV Reflective Panels aMong Congolese pregnAnt woMen Attending to Ante Natal Care Consultations
Brief Title: MAGIA H3S Point of Care Test Performance for HIV, HBV, HCV, and Syphilis Screening in Pregnant Women in DR Congo
Acronym: MAGICS MAM
Status: Not yet recruiting | Type: Observational
Sponsor: Gardiens de Vies (Other)
Collaborators: Institut Pasteur (Industry); MagIA Diagnostics (Industry)
Responsible Party: Principal Investigator, MAINDO ALONGO, Principal Investigator, Gardiens de Vies
Other Study IDs: 676/CNES/BN/PMMF/2025; 101159665 (Other Grant/Funding Number: Global Health EDCTP3)
Record Dates: First submitted 2026-01-07; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: HIV - Human Immunodeficiency Virus; HBV (Hepatitis B Virus); Hepatitis C Virus (HCV); Syphilis; Mother-to-Child Transmission; Performance; Point of Care STI Testing; TREAT B
Keywords: Triple elimination; Mother-to-child transmission; Democratic republic of the Congo
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis B; Hepatitis C; Syphilis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MAGIA H3S — MagiA H3S : Multiplex Point-of-Care test for the combined detection of Human Immunodeficiency Virus (HIV), Hepatitis B and C and Syphilis

SUMMARY:
Performance study to evaluate the clinical performance of the In-Vitro Diagnostic Medical Device MagIA H3S (a Multiplex Point-of-Care test for the combined detection of Human Immunodeficiency Virus (HIV), Hepatitis B and C and Syphilis) from pregnant women attending antenatal care (ANC) services in the Democratic Republic of the Congo. This study aligns with the WHO 2022-2030 strategy for the integrated elimination of mother-to-child transmission of HIV, HBV, HCV, and syphilis.

ELIGIBILITY:
Inclusion Criteria:

* Being pregnant, regardless of age or stage of pregnancy (prenatal period);
* Having signed an informed consent form at the start of prenatal care (CPN) to participate in the study.

Note: for pregnant minors, the consent of a parent or legal guardian is required;

* Have chosen to attend prenatal care at the healthcare facility selected for the study;
* Plan to give birth at the same healthcare facility where they were included in the study;
* Plan to attend postnatal care (PNC) and preschool consultations (PSC) at the same healthcare facility where they were included in the study.
* Plan to give birth at the same health facility where they were enrolled;
* Plan to attend postnatal consultations (PNC) and preschool consultations (PSC) at the same facility

Exclusion Criteria:

* Women in labor or who refuse to give their consent.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women attending antenatal care clinics among the 20 health facilities included for this study in DRCongo.
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-21 (Estimated)

PRIMARY OUTCOMES:
Performance evaluation of MagIA H3S in detection of HIV-Ab, HBAg, HCV-Ab and TP-Ab | Baseline
  Compare the sensitivity and specificity of the MAGIA H3S test with laboratory reference tests (ELISA/EIA for HIV, HBV and HCV, and syphilis) for detecting the following four markers in Congolese pregnant women: anti-HIV antibodies, anti-HCV antibodies, HBsAg and treponemal antibodies for syphilis.

SECONDARY OUTCOMES:
Positive predictive value (PPV) and negative predictive value (NPV) of MagiA H3S device | Baseline
  NPV and PPV calculated for each of the four diseases, using the laboratory tests as the reference for the entire population and according to different geographical area and socio-demographic context.
Sensitivity and specificity of MagiA H3S device to dignose HIV, HBV, HCV and syphilis. | Baseline
  For each of the four diagnoses, the Sensitivity and specificity of the MAGIA H3S will calculated and compared to the sensitivity and specificity of RDTs test, using fourth generation ELISA as the reference.
Stratum-specific sensitivity and specificity of the H3S test. | Baseline
  For each of the four diagnoses, the sensitivity and specificity of the MagIA H3S device will be calculated by stratifying them according to known infection and/or treatment history.
SE and SP, PPV and NPV of the MagIA TREATB test among pregnants women. | Up to 4 weeks
  Performance evaluation of MagiA TREATB test in detection of HbeAg, ALT and HbsAg quantification among pregnant women. The MagiA TREAT-B test that detect the Hbe-Ag, the ALT level and quantifies HbsAg will be compared to the laboratory tests as the reference.
Se and Sp of the MagIA TREAT-B test in postpartum women, 6 months after delivery | 6 month post partum
  Performance evaluation of MagiA TREATB test in detection of HbeAg, ALT and HbsAg quantification women who gave birth. The MagiA TREAT-B test that detect the Hbe-Ag, the ALT level and quantifies HbsAg will be compared to the laboratory tests as the reference.
Number and types of usage errors observed during the study as well as any malfunctions of the MagiA H3S device. | Baseline
Cotation of usability of the MagiA device from the users' perspective. | From baseline
  System usability scale will be used to assess the usability of use of the MagiA H3S test from healthcare personnel who have used the diagnostic tests. The score's scale ranges from 1 to 5. 1 means strongly disagree and 5 strongly agree.
Prevalence of HIV, hepatitis B and C viruses, and syphilis among pregnant women in the DRC. | Up to 4 weeks from baseline
  Prevalence of HIV, HBV, HCV and Syphilis using laboratory tests results of pregnant women in DRC.
Proportion of pregnant women who accepted the antenatal screening of HIV, HBV, HCV and Syphilis | Baseline
  The number of pregant women who accepted antenatal screening (rapid diagnostic tests and MagiA H3S) to detect HIV, HBV, HCV, and syphilis compared to total number of pregnant women attending antenatal services.
Proportion of positive results returned to pregnant women attending prenatal clinics in selected sites in the DRC. | Baseline
  Number of positive test results for HIV, HBV, HCV and Syphilis communicated to pregnant women who tested positive during antenatal consultations.
Cotation of Treatment adherence among positive pregnant women recieving treatment | Through study completion, an average of 2 year
  Treatment adherence of study participants receiving treatment will be assessed at each follow-up visit using the 8-item Morisky Medication Adherence Scale. The Morisky adherence scale yields a score ranging from 0 to 8, with higher scores indicating better adherence to treatment.
Proportion of vaccinated newborn born from positive HBV positive pregnants women within the first 24 hours. | At delivery
  Rate of newborns of pregnant women infected with HBV who received the hepatitis B vaccine
Rate of mother-to-child transmission for HIV, syphilis, HCV, and HBV. | Four to six weeks after birth for HIV, Six months after birth for HBV, at birth for syphilis and six weeks to tree months after birth for HCV post partum
  For each of the four infections: ratio between number of newborns born to positive pregnant women and number of positive newborns is calculated
Cost-effectiveness of the MAGIA H3S diagnostic test | Perioperative/Periprocedural
  Medical-economic evaluation of the MAGIA H3S diagnostic test by analyzing the costs associated with its implementation and its cost-effectiveness, compared to the absence of screening in routine antenatal care (status quo), and with the implementation of rapid HIV, HBV, HCV, and syphilis tests.
Cost-effectiveness of the MAGIA TREAT B diagnostic test to identify pregnant women eligible for antiviral prophylaxis against hepatitis B | Perioperative/Periprocedural
  * Total economic cost of introducing the MAGIA TREAT B test to identify pregnant women eligible for antiviral prophylaxis against Hepatitis B.
  * Cost-effectiveness assessment of the MAGIA TREAT B test, compared to the status quo and to viral load quantification or the HbeAg test.
Cost-effectiveness of the MAGIA TREAT B diagnostic test to identify women infected with hepatitis B virus who are eligible for long-term treatment for their own health | through study completion, an average of 2 years.
  * Total economic cost of introducing the MAGIA TREATB test to identify women infected with hepatitis B virus who are eligible for long-term treatment for their own health
  * Cost-effectiveness assessment of the MAGIA TREAT B test, compared to the status quo, as well as to the use of the APRI score, or the measurement of viral load and/or ALT levels.
Odds of pregnant women's preference regarding HBV diagnostic strategy for antenatal prophylaxis. | One month after inclusion
  Preference estimated as odd ratio from a discrete choice experiment.
Cotation of the capacity of health facilities to provide essential hepatitis care services | 1 to 2 months before the begining of the study
  Health facility service availability and readiness will be presented as percentage ranging from 0% to 100% for included indicators using the WHO's Service Availability and Readiness Assessment (SARA) tool. The study will describe the percentage of service availability and readiness for each health facility.

CONTACTS AND LOCATIONS:
Overall Officials: KANA LINGAMBU, MPH, Study Chair — Gardiens de Vies

IPD SHARING:
Plan to Share IPD: Yes
The IPD from this research will be shared upon written request by contacting the project coordinator, the president of MAGIA Diagnostics, and the study sponsor, the coordinator of GArdiens de Vies, at the following email addresses: paul.kauffmann@magia-diagnostics.com and olivier.kana@gardiensdevies.org
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From the end of the study up to 5 years later
Access Criteria: Researcher must write a request by contacting the project coordinator, the president of MAGIA Diagnostics, and the study sponsor, the coordinator of GArdiens de Vies, at the following email addresses: paul.kauffmann@magia-diagnostics.com and olivier.kana@gardiensdevies.org